CLINICAL TRIAL: NCT02633358
Title: Anti-inflammatory Effect of Therapeutic Hypothermia in Out-hospital Cardiac Arrest Patients With Cardiogenic Shock Via Interleukin-6 Trans-signaling
Brief Title: Anti-inflammatory Effect of Therapeutic Hypothermia in Out-hospital Cardiac Arrest Patients With Cardiogenic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH104-REC3-058
Record Dates: First submitted 2015-12-08; First posted 2015-12-17 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Arrest
Keywords: Acute myocardial infarction, cardiogenic shock
MeSH Terms: conditions — Heart Arrest; Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic hypothermia group (Experimental): Anti-inflammatory effect of therapeutic hypothermia. The hypothesis is anti-inflammatory effect triggered by IL-6 trans-signaling
  Interventions: Device: Therapeutic hypothermia group
- Control group (No Intervention): No therapeutic hypothermia for controlled data.

INTERVENTIONS:
Device: Therapeutic hypothermia group — Therapeutic hypothermia
  Arms: Therapeutic hypothermia group

SUMMARY:
Acute myocardial infarction complicated with cardiogenic shock trigger IL-6, the strong inflammatory response, result in multiple organ failure, even death.

While therapeutic hypothermia,to expect the possibility of anti-inflammatory effect via IL-6 bi-phasic effect and IL-10 , to improve the multiple organ failure, to increase survival rate and well cerebral performance.

DETAILED DESCRIPTION:
Despite emergency coronary revascularization coupled with medical stabilization, intra-aortic balloon pump have significantly improved survival in patients with cardiogenic shock complicating acute myocardial infarction, mortality still remains excessively high, being actually about 30-50%. Future research should focus on new therapeutic strategies, aimed to further decrease mortality rate of these patients or improve possible hospitalization and prognosis.

Heart pumping failure result in cardiogenic shock. Increased LA filling pressure result in acute pulmonary edema, hypoxemic respiratory failure, even congestive kidney and congestive liver. Decreased stroke volume result in hypoperfusion obviously direct induce acute renal failure, disturbance consciousness and lactate accumulation, even, shock liver. Multiple organ failure is the major mortality in the patients suffered from cardiogenic shock after acute myocardial infarction.

Cardiogenic shock remains the leading cause of death in patients hospitalized for myocardial infarction . Systemic inflammation , especially endovascular Interleukin-6, triggered by Tumor necrosis factor-alfa and Interleukin-1 beta result in inappropriate vasodilatation is observed in many patients with cardiogenic shock and may contribute to an excess mortality rate. In recent study, interleukin-6 represented a reliable independent early prognostic marker of 30-day mortality.

Therapeutic hypothermia (34℃) increase stroke volume, reduce muscle oxygen consumption and enhance anti-inflammatory action . The mechanism of anti-inflammatory effect for therapeutic hypothermia in cardiogenic shock is still unclear, need to further study in clinical trial. Furthermore, this study will provide new strategy to increase survival rate in cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-100 years
* Cardiogenic sock including initial lactate level >18 mg/dL, necessary of vasopressor to keep mean artery pressure >65mmHg after adequate fluid supply, and signs of reduced cardiac output including disturbance consciousness, cold limbs, decreased urine output, acute pulmonary congestion and so on.

Exclusion Criteria:

* Patient or family refuse
* Metastatic cancer
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-11-01; Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Da-Long Chen, Master, Study Director — Chnia Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitt KR, Tong G, Berger F. Mechanisms of hypothermia-induced cell protection in the brain. Mol Cell Pediatr. 2014 Dec;1(1):7. doi: 10.1186/s40348-014-0007-x. Epub 2014 Dec 1. PMID 26567101
- [Background] Bro-Jeppesen J, Kjaergaard J, Stammet P, Wise MP, Hovdenes J, Aneman A, Horn J, Devaux Y, Erlinge D, Gasche Y, Wanscher M, Cronberg T, Friberg H, Wetterslev J, Pellis T, Kuiper M, Nielsen N, Hassager C; TTM-Trial Investigators. Predictive value of interleukin-6 in post-cardiac arrest patients treated with targeted temperature management at 33 degrees C or 36 degrees C. Resuscitation. 2016 Jan;98:1-8. doi: 10.1016/j.resuscitation.2015.10.009. Epub 2015 Oct 23. PMID 26525271
- [Background] Forkmann M, Kolschmann S, Holzhauser L, Ibrahim K, Guenther M, Christoph M, Fuhrmann JT, Boscheri A, Schmeibetaer A, Strasser RH, Wunderlich C. Target temperature management of 33 degrees C exerts beneficial haemodynamic effects after out-of-hospital cardiac arrest. Acta Cardiol. 2015 Aug;70(4):451-9. doi: 10.1080/ac.70.4.3096893. PMID 26455248
- [Background] Nobile L, Lamanna I, Fontana V, Donadello K, Dell'anna AM, Creteur J, Vincent JL, Pappalardo F, Taccone FS. Greater temperature variability is not associated with a worse neurological outcome after cardiac arrest. Resuscitation. 2015 Nov;96:268-74. doi: 10.1016/j.resuscitation.2015.09.004. Epub 2015 Sep 16. PMID 26386374
- [Background] Bro-Jeppesen J, Kjaergaard J, Wanscher M, Nielsen N, Friberg H, Bjerre M, Hassager C. Systemic Inflammatory Response and Potential Prognostic Implications After Out-of-Hospital Cardiac Arrest: A Substudy of the Target Temperature Management Trial. Crit Care Med. 2015 Jun;43(6):1223-32. doi: 10.1097/CCM.0000000000000937. PMID 25756419
- [Background] Dankiewicz J, Nielsen N, Annborn M, Cronberg T, Erlinge D, Gasche Y, Hassager C, Kjaergaard J, Pellis T, Friberg H. Survival in patients without acute ST elevation after cardiac arrest and association with early coronary angiography: a post hoc analysis from the TTM trial. Intensive Care Med. 2015 May;41(5):856-64. doi: 10.1007/s00134-015-3735-z. Epub 2015 Mar 24. PMID 25800582
- [Derived] Chen D, Lin Y, Ko P, Lin J, Huang C, Wang G, Chang KC. Effect of targeted temperature management on systemic inflammatory responses after out-of-hospital cardiac arrest: A prospective cohort study. Medicine (Baltimore). 2024 Sep 20;103(38):e39780. doi: 10.1097/MD.0000000000039780. PMID 39312301
- [Derived] Chen DL, Chung CM, Wang GJ, Chang KC. Lactate-to-albumin ratio and cholesterol levels predict neurological outcome in cardiac arrest survivors. Am J Emerg Med. 2024 Sep;83:9-15. doi: 10.1016/j.ajem.2024.06.029. Epub 2024 Jun 25. PMID 38943710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2015 Jan. to 2018 Apr. Types of location: Cardiac intensive care units, China Medical University Hospital, Taichung, Taiwan
Groups:
- Therapeutic Hypothermia: Anti-inflammatory effect of therapeutic hypothermia. The hypothesis is anti-inflammatory effect triggered by IL-6 trans-signaling
  Therapeutic hypothermia: Therapeutic hypothermia
- Non-hypothermia: Control group for non-hypothermia. Anti-inflammatory effect of therapeutic hypothermia. The hypothesis is anti-inflammatory effect triggered by IL-6 trans-signaling
Period: Overall Study
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Started | 87 | 54
Completed | 87 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total 141 patients involved in this study. 87 patients divided in the therapeutic hypothermia group and 54 patients divided in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Hypothermia | Non-Hypothermia | Total
Number analyzed (Participants) | 87 | 54 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 30 | 80
  >=65 years | 37 | 24 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 70 | 42 | 112
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese in Taiwan | 86 | 54 | 140
  Japanese | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Taiwan | 87 | 54 | 141

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate - Number of Participants Alive
Description: Survival rate according to the number of participants alive in the 90 days after enrollment.
Time Frame: 90 days after enrollment
Population: Randomized divided to two groups including therapeutic hypothermia group and non-hypothermia group
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Number analyzed (Participants) | 87 | 54
Participants
  Survival | 55 | 20
  Non-survival | 32 | 34
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Non-hypothermia; Therapeutic hypothermia group compare with control group; Test type: Superiority — Therapeutic hypothermia need to have superiority in the survival rate after 90 days; p < 0.001, Chi-squared — P-value less than 0.05 means significant data; Test method for proportional data; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.41 to 0.82]

2. Secondary Outcome: Neurologic Outcome - Number of Participants
Description: Neurological outcome according to Cerebral performance Category scales: scales 1-2 in favor of favorable neurological outcome; scales 3-5 in favor of poor neurological outcome including severe cerebral disability, coma or vegetative state, brain death.
Time Frame: 90 days after enrollment
Population: Randomized divided to two groups including therapeutic hypothermia group and non-hypothermia group
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Number analyzed (Participants) | 87 | 54
Participants
  Favorable neurologic outcome | 30 | 10
  Poor neurologic outcome | 57 | 44
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Non-hypothermia; Therapeutic hypothermia group compare with control group; Test type: Superiority — Therapeutic hypothermia nee to have superiority in neurological outcome in the 90 days after enrollment; p = 0.04, Chi-squared — P value less than 0.05 means significant date; Test method for proportional data; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.66 to 0.98]

3. Other Pre Specified Outcome: Interleukin-6 - the Plasma Level of Participants
Description: IL-6 level change
Time Frame: between 6 and 24 hours after enrollment.
Population: Randomized divided to two groups including therapeutic hypothermia and non-hypothermia group
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Number analyzed (Participants) | 87 | 54
pg/mL
  6 hours after enrollment | 2064.1 (178.2) | 2392.4 (181.3)
  24 hours after enrollment | 914.5 (187.8) | 5125.0 (592.0)
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Non-hypothermia; Test type: Superiority; p < 0.05, t-test, 2 sided — P-value less than 0.05 is statistical significance

4. Other Pre Specified Outcome: Interleukin-6/Soluble Interleukin-6 Receptor Complex - the Plasma Level of Participants
Description: Interleukin-6/soluble Interleukin-6 receptor complex plasma level hint the pro-inflammatory pathway via Interleukin-6 trans-signaling
Time Frame: between 6 and 24 hours after enrollment
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Number analyzed (Participants) | 87 | 54
pg/mL
  6 hours after enrollment | 169.1 (7.6) | 188.1 (14.2)
  24 hours after enrollment | 207.8 (14.6) | 319.7 (24.5)
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Non-hypothermia; Test type: Superiority; p < 0.05, t-test, 2 sided — P-value less than 0.05 is statistical significance

5. Other Pre Specified Outcome: Soluble Interleukin-6 Receptor - the Plasma Level of Participants
Description: Check the soluble Interleukin-6 plasma level at 6 hours and 24 hours after enrollment
Time Frame: between 6 and 24 hours after enrollment
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Therapeutic Hypothermia | Non-hypothermia
Number analyzed (Participants) | 87 | 54
ng/mL
  6 hours after enrollment | 40.6 (1.6) | 37.9 (1.6)
  24 hours after enrollment | 37.9 (1.3) | 35.7 (1.5)
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Non-hypothermia; Test type: Superiority; p < 0.05, t-test, 2 sided — P-value less then 0.05 is statistical significance

ADVERSE EVENTS:
Time Frame: 90-day follow up
Groups:
- Therapeutic Hypothermia; Non-Hypothermia: Adverse events including ventricular arrhythmia, active bleeding, death due to lower core temperature less than 32 degree Celsius.
Arm/Group | Therapeutic Hypothermia | Non-Hypothermia
All-Cause Mortality (participants affected / at risk) | 32/87 | 34/54
Serious Adverse Events (participants affected / at risk) | 57/87 | 44/54
Other Adverse Events (participants affected / at risk) | 0/87 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Hypothermia (N=87) | Non-Hypothermia (N=54)
Severe cerebral disability (Nervous system disorders) | 11 (11) | 4 (4) — Severe cerebral disability
Coma or vegetative state (Nervous system disorders) | 14 (14) | 6 (6) — Coma or vegetative state
Brain death (Nervous system disorders) | 32 (32) | 34 (34) — Brain death

LIMITATIONS AND CAVEATS:
Pregnancy, terminal and metastatic cancer, uncontrolled bleeding and family refuse inform consent had been excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT02633358/Prot_SAP_000.pdf